CLINICAL TRIAL: NCT01149187
Title: Usefulness of Interferon-gamma Release Assay in Diagnosing Pulmonary Nodules
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Young Whan Kim/professor, Seoul National University Hospital
Other Study IDs: SeoulNUH-IGRA-01
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Solitary Pulmonary Nodule
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — the investigaters will use the whole blood sample for interferon-gamma release assay.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IGRA in solitary pulmonary nodules: Inpatients who undergo percutaneous needle biopsy for diagnosis of pulmonary nodules in Seoul National University hospital for six months are going to be included. Patients who are not tolerable for PCNB or do not agree the enrollment of study will be excluded.

SUMMARY:
Among the causes of the solitary pulmonary nodule (SPN), benign causes including tuberculosis was noted on 15 to 60 percents in various studies.

Although the characteristics of chest imaging is helpful in diagnosis and percutaneous needle biopsy for pulmonary nodule has been represented high diagnostic yield in many reports, but still surgical biopsy has been needed in definite diagnosis of pulmonary nodules in many cases.

The aim of this study is to evaluate the usefulness of interferon-gamma release assay in addition to the percutaneous needle biopsy, in diagnosis of pulmonary nodules.

DETAILED DESCRIPTION:
Among the patients who failed to diagnosis by percutaneous needle biopsy and needed to have Surgical biopsy, thirty percents of the patients were diagnosed as benign nodules and about six percents were diagnosed as tuberculosis in Seoul National University Hospital during 2007-2008.

The investigators want to know whether conducting an interferon-gamma release assay in addition to percutaneous needle biopsy is helpful in diagnosis of lung nodules.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* in patients with solitary pulmonary nodule
* who had percutaneous needle biopsy for diagnosis of lung nodule

Exclusion Criteria:

* patients who do not agree the study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among the inpatients who got percutaneous needle biopsy for pulmonary nodule during the study periods are going to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Positive rate of the interferon-gamma release assay | within 36hrs after blood sampling
  the result of the interferon-gamma release assay is reported in three different categories as positive, negative or indeterminate. We want to know whether the positive rate of the interferon-gamma release asssay would be significantly different according to the pathologic diagnosis of lung nodules confirmed by percutaneous needle biopsy.

SECONDARY OUTCOMES:
Positive rate of the Tuberculin skin test | 48hours after tuberculin skin test
  We will conduct Tuberculin skin test and evaluate the whether the positive rate of the Tuberculin skin test would be different according to the pathologic diagnosis of lung nodules confirmed by percutaneous needle biopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Young Whan Kim, Seoul, South Korea